CLINICAL TRIAL: NCT01639586
Title: Comparaison du Service Rendu à la Personne Atteinte d'Une Maladie d'Alzheimer et de l'Aidant Par Trois Types de Prises en Charge (Plateforme, Accueil de Jour et Groupe contrôle
Brief Title: Comparison for the Patient With Alzheimer Disease the Impact of Three Different Groups of Patient Care
Acronym: COMPARSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Clinical Research and Innovation (Other)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Department of Clinical Research and Innovation (drc), Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-A00167-34
Record Dates: First submitted 2012-03-23; First posted 2012-07-12 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Day Care, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- D (Active Comparator): Impact of the day care on health profit of patient
  Interventions: Behavioral: Day care
- C (Active Comparator): No access to a respite structure
  Interventions: Behavioral: No access to a respite structure
- B (Active Comparator): Respite platform
  Interventions: Behavioral: respite platform

INTERVENTIONS:
Behavioral: respite platform — Impact of the respite platform patient care on health profit
  Arms: B
Behavioral: Day care — Impact of the day care on health profit of patient
  Arms: D
Behavioral: No access to a respite structure — Control group without access to a respite structure
  Arms: C

SUMMARY:
One of the interests of the Alzheimer Plan 2008-2010 is to provide increase support to helping families. It's also of major to involve the patient in the most active treatment possible, encouraging social inter relationship as well as cognitive and behavioural stimulation activities.

In the frame of non drug related approaches to Alzheimer disease (AD), several research projects and actions have already been conducted, but no specific study concerning the efficiency of different types of respite care structures have been conducted so far in France. The present project concerns the thematic of the frame "Development and diversification of respite care structures".

A platform is defined in the Alzheimer Plan as a "diversified range of despite structures according to patients' needs and informal caregivers' expectations" providing several objectives:

Two objectives targeting the informal caregivers:

* offer spare time or tutored
* inform, support and accompany

Two objectives targeting the patients:

* encourage maintain of the patient social life and relationships and work together towards his/her psychological and emotional well-being
* contribute to improve functional cognitive and sensory capacities

The study COMPARSE suggests to compare for the patient - informal caregiver couple, the impact of three different groups of patient care on health profit; resit platform (P), the day care group (D), the control group without access to a respite structure (C).

ELIGIBILITY:
Inclusion criteria

* patient affect by Alzheimer disease or related pathology
* patient with an informal caregiver
* patient not using any respite structure
* signed informed consent (patient and informal caregiver)
* affiliate to social security

Exclusion criteria

* patient without informal caregiver
* patient include in another clinical protocol

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Analysis of the perceived and diagnosed health evolution of the patient | at baseline, one month and nine month
  Realize neuropsychological evaluation and satisfaction degree evaluation of the patient and the informal caregiver to compare different types of respite care structures

SECONDARY OUTCOMES:
Efficacity of the different structures | at baseline, one month and nine month
  Assess autonomy level of patient Realize sociological qualitative analysis and economic evaluation by comparing differents structures

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pradier, PHD MD, Principal Investigator — Département de Santé Publique - CHU de Nice
Locations (1):
- Le Duff, Nice, France